CLINICAL TRIAL: NCT02939937
Title: a Phase II Double Blind, Randomized, Placebo Controlled Trial of Effect of Phenytoin on the Ganglion Cell Inner Plexiform Layer (GCIPL) Thickness and Visual Field in Patients With a First Episode of Acute Optic Neuritis
Brief Title: Effect of Phenytoin on the Ganglion Cell Layer in Patients With Optic Neuritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9411257013
Record Dates: First submitted 2016-08-08; First posted 2016-10-20 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2018-04

CONDITIONS: Optic Neuritis
MeSH Terms: conditions — Optic Neuritis | interventions — Phenytoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: participant , investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phenytoin (Experimental): patients received phenytoin 100mg three time daily up to 3 months
  Interventions: Drug: Phenytoin
- placebo (Experimental): patients received placebo 100 mg three time daily for 3 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Phenytoin — 100 mg phenytoin three time daily for three months, and phenytoin levels will be taken at one and three months later.
  Other Names: epanutin
  Arms: phenytoin
Drug: placebo — 100 mg placebo three time daily for three months, and phenytoin levels will be taken at one and three months later.
  Arms: placebo

SUMMARY:
Optic neuritis typically occurs in young (mean age, 32 years), female (77%) patients, and it presents as subacute monocular visual loss that develops over several days.

As yet, treatment with intravenous corticosteroid for optic neuritis had no long-term beneficial effect on vision.

There are a number of factors that contribute to nerve fibre damage including increased level of sodium, so blocking sodium entry could help to protect them against damage.

The main objective of the study is determine whether phenytoin (which blocks sodium entry) can protect nerve fibre and improve final visual function after optic neuritis.

ELIGIBILITY:
Inclusion Criteria:

* isolated, unilateral, first acute optic neuritis (confirmed by neuroophthalmologist)
* willing to receive a steroidal regimen
* no pathologic finding in first oct
* no pathology and history of optic neuritis in contralateral eye
* <14 days since onset visual loss

Exclusion Criteria:

* Contraindication or known allergy to Phenytoin
* Use of a calcium channel or sodium channel blocker in the past 2 months
* Corticosteroid use in the past 2 months
* Pregnancy
* Significant cardiac, renal or liver abnormalities
* Prior clinical episode of optic neuritis in either eye
* Bilateral acute optic neuritis
* Known ocular or neurological conditions or abnormalities other than refractive error that impair visual function
* Refractive error of greater than +5 or -5 diopters
* Any condition that may interfere with performance of Optical Coherence Tomography (OCT): corneal, lens or fundoscopic abnormality, a co-morbid ocular condition not related to optic neuritis as detected on the OCT reading

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2019-01-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Research Center Farabi Hosoital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phenytoin | Placebo
Started | 21 (5 patients had drug reaction and 1 patient excluded from study,) | 50 (3 patients excluded from study)
Completed | 15 | 47
Not Completed | 6 | 3
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenytoin | Placebo | Total
Number analyzed (Participants) | 21 | 50 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 50 | 71
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 40 | 54
  Male | 7 | 10 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: 6 subjects in phenytoin group and 3 subjects in placebo group were excluded from our study and this left 15 patients in phenytoin and 47 subjects in placebo group to be analysed.
  participants
    Iran: number analyzed (Participants) | 15 | 47 | 62
    Iran | 15 | 47 | 62

OUTCOME MEASURES:

1. Primary Outcome: Retinal Ganglion Cell Inner Plexiform Layer Thickness
Description: ganglion cell inner plexiform layer thickness measure in 8 sectors by Heidelberg spectral-domain Optical Coherence Tomography
Time Frame: Measured at baseline and month 1, 6
Population: incomplete follow up from baseline to 6 month
Measure: Mean (Standard Deviation); unit: micron
Arm/Group | Phenytoin | Placebo
Number analyzed (Participants) | 15 | 47
micron
  baseline | 36.56 (6.61) | 34.65 (8.49)
  1 month: number analyzed (Participants) | 12 | 28
  1 month | 31 (6.61) | 29.42 (5.98)
  6 months: number analyzed (Participants) | 11 | 26
  6 months | 30.70 (5.56) | 32.12 (9.10)

2. Primary Outcome: Macular Layer Thickness
Description: macular layer thickness measure in 8 sectors by Heidelberg spectral domain Optical Coherence Tomography
Time Frame: Measured at baseline and month 1, 6
Population: incomplete follow up
Measure: Mean (Standard Deviation); unit: micron
Arm/Group | Phenytoin | Placebo
Number analyzed (Participants) | 15 | 47
micron
  baseline | 262.73 (22.02) | 265.98 (22.5)
  1 month: number analyzed (Participants) | 11 | 28
  1 month | 255 (19.72) | 264.39 (22.53)
  6 months: number analyzed (Participants) | 11 | 26
  6 months | 269 (28.29) | 268.37 (22.69)

3. Primary Outcome: Best Corrected Visual Acuity
Description: Best corrected visual acuity is converted to logMAR (logarithms of minimum angle of resolution) by statistical calculation.
Time Frame: at baseline and month 6
Population: incomplete follow up
Measure: Mean (Standard Deviation); unit: log mar
Arm/Group | Phenytoin | Placebo
Number analyzed (Participants) | 15 | 47
log mar
  baseline | 1.44 (0.98) | 1 (0.83)
  6 months: number analyzed (Participants) | 11 | 26
  6 months | 0.04 (0.067) | 0.13 (0.448)

4. Primary Outcome: Visual Field Mean Deviation in Decibel
Description: The visual field is performed by the Swedish interactive thresholding algorithm standard 24-2 perimeter (Carl Zeiss mediated, Dublin, California).
Time Frame: Measured at baseline and month 6
Population: incomplete follow up
Measure: Mean (Standard Deviation); unit: db
Arm/Group | Phenytoin | Placebo
Number analyzed (Participants) | 15 | 47
db
  Baseline visual field mean deviation (MD) | -17.07 (11.41) | -17.76 (11.81)
  6 months MD: number analyzed (Participants) | 11 | 26
  6 months MD | -3.89 (4.46) | -5.16 (7.49)

5. Secondary Outcome: Retinal Nerve Fibre Layer Thickness in Micrometer
Description: Retinal nerve fibre layer thickness measure in 8 sectors by Heidelberg spectral-domain Optical Coherence Tomography
Time Frame: Measured at baseline and month1 ,6
Population: incomplete follow up
Measure: Mean (Standard Deviation); unit: micron
Arm/Group | Phenytoin | Placebo
Number analyzed (Participants) | 15 | 47
micron
  Baseline | 131.8 (36.56) | 124.87 (47.51)
  1 month: number analyzed (Participants) | 13 | 28
  1 month | 93.85 (8.64) | 97.41 (23)
  6 months: number analyzed (Participants) | 11 | 26
  6 months | 77.7 (20.03) | 78.61 (18.97)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Phenytoin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/50
Other Adverse Events (participants affected / at risk) | 4/21 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenytoin (N=21) | Placebo (N=50)
steven johnson (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — steven johnson syn,Stevens-Johnson syndrome (SJS) is a type of severe skin reaction
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenytoin (N=21) | Placebo (N=50)
skin reaction (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) — sever skin reaction to drug except sjs

LIMITATIONS AND CAVEATS:
1. Shorter follow up
2. Poor compliance for oral drug intake

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-04-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT02939937/Prot_000.pdf
  • Informed Consent Form (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT02939937/ICF_001.pdf
  • Statistical Analysis Plan (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT02939937/SAP_002.pdf